CLINICAL TRIAL: NCT04525872
Title: Parenteral Nutrition Light Protection and Premature Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-00378
Record Dates: First submitted 2020-07-24; First posted 2020-08-25 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth | interventions — Lipids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Premature infants (Experimental): Premature infants who are expected to receive TPN for a minimum of 5 days and infants with gastrointestinal surgical problems (e.g., ileal atresia, gastroschisis), expected to receive TPN for a minimum of 5 days
  Interventions: Other: Full parenteral nutrition light protection of the bag, tubing and lipids

INTERVENTIONS:
Other: Full parenteral nutrition light protection of the bag, tubing and lipids — Each infant enrolled in this study will receive full PN light protection including the PN bag, lipids and tubing.

SUMMARY:
Investigators propose a prospective study to investigate the effect of full light protection of the PN on cholestasis and other oxidative stress associated diseases in premature infants when they receive PN for more than one week. Each infant enrolled in this study will receive full PN light protection including the PN bag, lipids and tubing. Demographic characteristics, clinical outcomes (incidence of cholestasis, feeding tolerance, BPD, ROP, NEC and mortality) and oxidative stress markers (e.g., carboxyhemeglobin) will be evaluated. Phase one of this study employed a retrospective chart review methodology to evaluate the effect of no PN light protection vs partial PN light protection (PN solution only while it's the tubing and lipids remained exposed to light). Infants from phase one of this study will serve as the controls in the evaluation the effect of full PN light protection on the cholestasis, clinical outcomes and oxidative stress. Investigators propose to collect urine and saliva samples in infants who we expect to receive PN for a minimum of 5 days, on days 0, 3, 5 and every 7 days after TPN initiation until 2 weeks after the end of IV nutrition to evaluate oxidative stress.

ELIGIBILITY:
Inclusion criteria

* Preterm infants <32 weeks of gestation, who receive TPN for a minimum of 5 days
* Infants with gastrointestinal surgical problems (e.g., ileal atresia, gastroschisis), expected to receive TPN for a minimum of 5 days Exclusion criteria
* Infants who receive TPN for <5 days
* Infants who developed cholestasis due to non-TPN-related causes

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Serum levels of direct bilirubin | Baseline, 2 weeks after the end of IV nutrition
  Change from baseline
Serum levels of liver enzymes | Baseline, 2 weeks after the end of IV nutrition
  Change from baseline
Serum levels of triglycerides | Baseline, 2 weeks after the end of IV nutrition
  Change from baseline
Serum levels of carnitine | Baseline, 2 weeks after the end of IV nutrition
  Change from baseline
Serum levels of total bilirubin | Baseline, 2 weeks after the end of IV nutrition
  Change from baseline

SECONDARY OUTCOMES:
Oxidative stress | Baseline, 2 weeks after the end of IV nutrition
  Change from baseline
Incidence of bronchopulmonary disease (BPD) | Days 0, 3, 5, and every 7 days after TPN initiation until 2 weeks after the end of IV nutrition
Incidence of retinopathy of prematurity (ROP) | Days 0, 3, 5, and every 7 days after TPN initiation until 2 weeks after the end of IV nutrition
Incidence of necrotizing enterocolitis (NEC) | Days 0, 3, 5, and every 7 days after TPN initiation until 2 weeks after the end of IV nutrition
Mortality | Days 0, 3, 5, and every 7 days after TPN initiation until 2 weeks after the end of IV nutrition

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Tiozza, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: caterina.tiozzo@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to caterina.tiozzo@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.